CLINICAL TRIAL: NCT00916045
Title: Pilot Study of Unrelated Cord Blood Transplantation in Patients With Poor Risk Haematological Malignancies
Brief Title: Pilot Study of Unrelated Cord Blood Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Recruitment issues
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Dr Antonio Pagliuca, King's College Hospital NHS Foundation Trust
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07CC12; REC - 07/H0808/193; EudraCT - 2007-001657-26
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2012-03

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Lymphoblastic, Acute; Lymphoma, Non-Hodgkin; Hodgkin Disease; Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Non-Hodgkin; Hodgkin Disease; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Thiotepa; fludarabine; Busulfan; thymoglobulin; Cyclosporine; Mycophenolic Acid; Cyclophosphamide; Radiotherapy; Melphalan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Myeloblative conditioning regimen (Other)
  Interventions: Drug: Thiotepa; Drug: Fludarabine; Drug: Intravenous busulphan; Drug: Thymoglobulin; Drug: Ciclosporin; Drug: Mycophenolate mofetil (MMF)
- Reduced intensity conditioning regimen - FluCyTBI (Other)
  Interventions: Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Radiotherapy; Drug: Thymoglobulin; Drug: Ciclosporin; Drug: Mycophenolate mofetil (MMF)
- Reduced intensity conditioning regimen - FluMel (Other)
  Interventions: Drug: Fludarabine; Drug: Melphalan; Drug: Thymoglobulin; Drug: Ciclosporin; Drug: Mycophenolate mofetil (MMF)

INTERVENTIONS:
Drug: Thiotepa
  Arms: Myeloblative conditioning regimen
Drug: Fludarabine
  Arms: Myeloblative conditioning regimen
Drug: Intravenous busulphan
  Other Names: Busilvex
  Arms: Myeloblative conditioning regimen
Drug: Thymoglobulin
  Arms: Myeloblative conditioning regimen
Drug: Ciclosporin
  Arms: Myeloblative conditioning regimen
Drug: Mycophenolate mofetil (MMF)
  Arms: Myeloblative conditioning regimen
Drug: Fludarabine
  Arms: Reduced intensity conditioning regimen - FluCyTBI
Drug: Cyclophosphamide
  Arms: Reduced intensity conditioning regimen - FluCyTBI
Radiation: Radiotherapy
  Arms: Reduced intensity conditioning regimen - FluCyTBI
Drug: Thymoglobulin
  Arms: Reduced intensity conditioning regimen - FluCyTBI
Drug: Ciclosporin
  Arms: Reduced intensity conditioning regimen - FluCyTBI
Drug: Mycophenolate mofetil (MMF)
  Arms: Reduced intensity conditioning regimen - FluCyTBI
Drug: Fludarabine
  Arms: Reduced intensity conditioning regimen - FluMel
Drug: Melphalan
  Arms: Reduced intensity conditioning regimen - FluMel
Drug: Thymoglobulin
  Arms: Reduced intensity conditioning regimen - FluMel
Drug: Ciclosporin
  Arms: Reduced intensity conditioning regimen - FluMel
Drug: Mycophenolate mofetil (MMF)
  Arms: Reduced intensity conditioning regimen - FluMel

SUMMARY:
The purpose of this study is to determine the safety and feasibility of unrelated double and single cord blood transplantation in patients with haematological malignancies using reduced-intensity or myeloablative conditioning regimens.

ELIGIBILITY:
DISEASE INCLUSION CRITERIA:

In general this encompasses all haematological disorders where a volunteer unrelated donor transplant is clinically indicated.

1. Acute, chronic leukaemia or myelodysplastic syndrome for which allogeneic transplantation is considered as the best treatment option.

   1. Acute myeloid leukaemia (AML) in first complete remission (CR1) with one of the following characteristics:

      * High risk cytogenetic or molecular alterations (e.g. t(9;22), deletion 7/7q-, monosomy 5 or del(5q), 3q26 alterations, complex karyotype [3 or more anomalies], p53 alterations, 11q23 especially t(6;11) abnormalities, FLT-3 ITD)
      * Leukocytes at diagnosis > 50 x109/l (except in cases with good prognosis molecular rearrangements for which leukocytes should be > 100 x 109/l)
   2. Myelodysplastic syndromes

      * International Prognosis Index (IPSS) above 1 (intermediate group 2 or high risk)
      * IPSS 0 or 0.5 in the presence of cytopenias requiring treatment.
   3. Therapy related AML or MDS in first CR
   4. AML or MDS in second (CR2) or subsequent CR
   5. Ph'-positive chronic myeloid leukaemia

   i. In first chronic phase if refractory and/or intolerance to tyrosine kinase inhibitors is clearly demonstrated ii. In second chronic phase
2. Acute lymphoblastic leukaemia (ALL)

   a. In CR1 with one of the following characteristics: i. Very high risk chromosome or molecular alterations (e.g. t(9;22), t(4;11), complex karyotype in adults, bcr/abl rearrangements, MLL rearrangements) ii. Slow response to induction treatment defined as the presence of >10% blasts in bone marrow at day 14 of induction treatment iii. Adults aged > 30 years iv. Adults with B ALL cell line with a number of leukocytes at diagnosis >25 x 109/L or T ALL cell line with a number of leukocytes at diagnosis >100X109/L

   b. In CR2 or subsequent CR
3. Non-Hodgkin's lymphoma

   1. Follicular NHL: in second or subsequent complete or partial remission
   2. Mantle cell NHL: in second or subsequent complete or partial remission
   3. High grade NHL: in second complete or very good partial remission
4. Hodgkin's disease

   a. in second or subsequent complete or partial remission
5. Chronic lymphocytic leukaemia.

   1. in second or subsequent remission
   2. with adverse risk prognostic features in first remission
6. Acquired bone marrow failure syndromes
7. Other haematological malignancies for which UD bone marrow transplantation is indicated

PATIENT SELECTION

Inclusion criteria: myeloablative conditioning regimen

1. Aged under 35 years and greater than 18 years
2. Absence of HLA compatible related donor.
3. Need for an urgent transplantation or absence of HLA-compatible VUD after searching the international registries.
4. Patients with a HLA-compatible VUD but whose donor is considered by the transplantation centre as unsuitable will also be eligible.
5. Availability of suitable UD-UCB unit/s.
6. Informed consent.

Exclusion criteria: myeloablative conditioning regimen

1. Patients with an available 5-6/6 HLA-A, -B, -DRB1 matched sibling donor or 10/10 unrelated bone marrow donor
2. ECOG performance status worse than 2
3. Cardiac insufficiency requiring treatment, symptomatic coronary artery disease or LVEF less than 40%.
4. Hepatic disease, with total bilirubin above 20umol/l or AST > 3 times upper limit of normal.
5. Severe hypoxaemia, pO2 < 70 mm Hg, with decreased DLCO < 70% of predicted; or mild hypoxemia, pO2 < 80 mm Hg with severely decreased DLCO < 60% of predicted.
6. Impaired renal function (creatinine > 2 times upper limit of normal or creatinine clearance < 50% for age, gender, weight).
7. Patients who have received previous treatment with Thymoglobulin®
8. HIV or HTLV positive patients.
9. Female patients who are pregnant or breast feeding due to risks to foetus from conditioning regimen and potential risks to nursing infants.
10. Life expectancy severely limited by diseases other than the disease indication for transplant
11. Serious concurrent untreated infection e.g. active tuberculosis, mycoses or viral infection
12. Serious psychiatric/ psychological disorders
13. Absence of /inability to provide informed consent
14. Serious diseases that prevent treatments with chemotherapy
15. Myelofibrosis

Inclusion criteria: reduced-intensity conditioning regimen (For both FluMel & FluCyTBI regimens):

1. Age under 70 years and older than 18 years
2. Absence of HLA compatible related donor.
3. Need for an urgent transplantation or absence of HLA-compatible VUD after searching the international registries.
4. Patients with a HLA-compatible VUD but whose donor is considered by the transplantation centre as unsuitable will also be eligible.
5. Availability of suitable UD-UCB unit/s.
6. Informed consent.

Exclusion Criteria: reduced-intensity conditioning regimen (For both FluMel & FluCyTBI regimens):

1. Patients with an available 5-6/6 HLA-A, -B, -DRB1 matched sibling donor or 10/10 unrelated bone marrow donor
2. ECOG performance status worse than 2
3. Cardiac insufficiency requiring treatment, symptomatic coronary artery disease or LVEF less than 35%.
4. Hepatic disease, with total bilirubin greater than 2 times upper limit of normal or AST > 5 times upper limit of normal.
5. Severe hypoxaemia, pO2 < 70 mm Hg, with decreased DLCO < 50% of predicted; or mild hypoxemia, pO2 < 80 mm Hg with severely decreased DLCO < 50% of predicted.
6. Impaired renal function (creatinine > 2 times upper limit of normal or creatinine clearance < 50% for age, gender, weight).
7. Previous irradiation that precludes the safe administration of an additional dose of 200 cGy of total body irradiation (TBI).
8. Patients who have received previous treatment with Thymoglobulin®
9. HIV or HTLV positive patients.
10. Female patients who are pregnant or breast feeding due to risks to foetus from conditioning regimen and potential risks to nursing infants.
11. Life expectancy severely limited by diseases other than the disease indication for transplant
12. Serious concurrent uncontrolled infection e.g. active tuberculosis, mycoses or viral infection
13. Serious psychiatric/ psychological disorders
14. Absence of /inability to provide informed consent
15. Within 6 months of prior myeloablative transplant.
16. Patients with acute leukaemia in morphological relapse/ persistent/ progressive disease
17. Intermediate or high grade NHL, mantle cell NHL and Hodgkin's disease that is refractory or progressive on salvage therapy.
18. Myelofibrosis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Treatment related mortality at day 100 | Day 100

SECONDARY OUTCOMES:
Disease free survival at one year post-transplant for each cohort | 1 year
Chimerism | Days 14 (myeloblative conditioning only), 28, 56, 100 and months 6 and 12
Incidence of neutrophil engraftment by day 42 | Days 14, 28 and 42
Incidence of platelet engraftment by 6 months | Days 14, 28, 56, 100 and month 6
Incidence of grade II-IV and III-IV acute GVHD | Days 28, 56, 100 and months 6, 9, 12, 18 and 24
Incidence of chronic GVHD during the first year | Day 100 and months 6 and 12
One year overall survival for each treatment cohort | 1 year
Incidence of systemic infections | Twice a week pre-transplant to day 100 then weekly or as clinically indicated
Incidence of CMV, adenovirus and EBV activation | Twice a week pre-transplant to day 100 then weekly or as clinically indicated
Immune reconstitution | Days 14, 28, 56, 100 and months 6, 9, 12, 18 and 24
Dynamics of EBV infection and immunity following cord blood transplantation | Days 14, 28, 56, 100 and months 6, 9 and 12
The development (if any) of transplant associated post transplant lymphoproliferative disease (PTLD) | Days 14, 28, 56, 100 and months 6, 9 and 12
Identify any possible predictive markers for patients most at risk of PTLD development | Days 14, 28, 56, 100 and months 6, 9 and 12
Quality of life | Pre-transplant and months 6, 12, 18 and 24
Incidence of one year relapse or disease progression for each treatment cohort | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pagliuca, MBBS, MA, FRCP, FRCPath, Principal Investigator — King's College Hospital NHS Trust
Locations (1):
- King's College Hosptial NHS Foundation Trust, London, United Kingdom